CLINICAL TRIAL: NCT02659085
Title: A Randomized Controlled Non-inferiority Trial Comparing Ketamine With ECT in Patients With Major Depressive Disorder
Brief Title: Ketamine as an Alternative Treatment to ECT in Major Depressive Disorder
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Pouya Movahed Rad (Other)
Responsible Party: Sponsor-Investigator, Pouya Movahed Rad, MD, PhD, Region Skane
Organization: Region Skane (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2011-001520-37
Record Dates: First submitted 2015-12-07; First posted 2016-01-20 (Estimated); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Depressive Disorder, Major
Keywords: Depressive Disorder, Major; Antidepressive Agents/adverse effects; Depressive Disorder, Major/drug therapy; Infusions, Intravenous; Ketamine/administration & dosage*; Ketamine/adverse effects; Treatment Outcome; Electroconvulsive therapy
MeSH Terms: conditions — Depressive Disorder, Major; Depressive Disorder | interventions — Ketamine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Electroconvulsive Therapy (ECT) (Active Comparator): ECT given in line with standard procedures (including anesthesia, muscle relaxation and oxygenation) thrice weekly. Each participating clinic decides for each patient whether the treatment is given uni- or bilateral, as well as the exact stimulation parameters. Choice of anesthetic drug (e.g. thiopental of propofol) and muscle relaxant is done by local anesthesiologist. The procedure differs in no way from how a given patient would have been treated if he or she were not included in the study.
  Interventions: Procedure: ECT
- Ketamine IV Infusion (Experimental): Ketamin intra venous infusions of racemic ketamine (0.5mg/kg), delivered over a period of 40 minutes thrice weekly, as ECT (Monday, Wednesday and Friday).
  Interventions: Drug: Ketamine IV Infusion

INTERVENTIONS:
Drug: Ketamine IV Infusion — Patients randomized to the experimental treatment receive intravenous infusions of racemic ketamine (0.5 mg/kg), delivered over a period of forty minutes thrice weekly (Monday, Wednesday, Friday) under supervision.
  Other Names: Ketamine
  Arms: Ketamine IV Infusion
Procedure: ECT — ECT given in line with standard procedures (including anesthesia, muscle relaxation and oxygenation) thrice weekly.
  Arms: Electroconvulsive Therapy (ECT)

SUMMARY:
Developing more effective and faster acting antidepressant is of outmost clinical importance. Available antidepressant therapies have a delayed therapeutic effect. It typically takes several weeks before symptom relief is evident. Furthermore, antidepressants are relatively ineffective - as many as 30% of patients do not respond to any medication at all. In this study the investigators evaluate the NMDA-receptor antagonist ketamine as a potentially new antidepressant treatment for severely depressed patients and compare its effectiveness with that of electroconvulsive therapy (ECT).

DETAILED DESCRIPTION:
In line with the PICO model, patient selection and procedures for experimental and control treatments and outcome measures are rigorously defined. Inpatients, aged 18-85, diagnosed with major depressive disorder (MDD, according to DSM-IV), that have been offered and have accepted ECT, are eligible to participate. Patients must be proficient in spoken and written Swedish, and score ≥ 20 points on the Montgomery Åsberg Depression Rating Scale (MADRS). Exclusion criteria are known allergy to the active substance; co-morbid conditions that could interfere with the treatment (e.g. primary psychosis); habitual difficulties to speak, hear, remember or reason; on-going or recent (6 months) drug abuse; treatment according to LPT (Lagen om psykiatrisk tvångsvård; Compulsory Psychiatric Care Act); and a number of cardiovascular conditions.

Patients randomized to the experimental treatment receive intravenous infusions of racemic ketamine (0.5 mg/kg), delivered over a period of forty minutes thrice weekly (Monday, Wednesday, Friday). Patients in the control group receive ECT in line with standard procedures (including anesthesia, muscle relaxation and oxygenation) thrice weekly. ECT was chosen as the reference treatment as it is the most effective treatment for patients suffering from moderate to severe depression.

Primary outcome is the proportion of patients in remission after 4 weeks of treatment in each arm. Remission is defined as a MADRS ≤ 10.

The study uses a non-inferiority design. Demonstrating superiority of ketamine was not an option based on the number of patients needed to gain sufficient power with such a design. Also, the investigators do not believe that ketamine treatment needs to be more effective, at least not in terms of the primary outcome. ECT is associated with side effects (in particular amnesia during the treatment period, but some patients also report persistent memory problems) and patients need to be anaesthetised under the supervision of a anaesthesiologist. The treatment is thus fairly demanding and expensive. A significant amount of patients are also unwilling to undergo ECT. Given non- inferiority of ketamine regarding the primary outcome, and given that it is associated with fewer side effects or shorter time to remission and does not involve the need for anaesthesia, in a risk-benefit analysis the scale might be tipped in favour of ketamine, even if it is not superior per se.

Secondary outcomes include proportion of patients in re mission and /or response and symptomatic relief at follow-up time points (3, 6 and 12 months after treatment cessation). Also addressed is how the two treatments affect cognition. A computerized test battery, the Cambridge Automated Neuropsychological Test Automated Battery (CANTAB) is administered prior to the first treatment, after two weeks, shortly after remission and at three additional time points (3, 6 and 12 months) after conclusion of the treatment. See figure for specification and description of cognitive tests.

Blood samples are drawn before the first treatment and 2-3 months after finishing treatment. Apart from plasma and serum samples (which will be used for later analysis of potential biomarkers such as IL 6 and D-serine), additional blood is collected for genomic DNA analysis. A total of 4 x 6 mL are taken at each occasion. Blood samples are stored at the regional biobank.

Time to response will be analysed with parametric survival analysis (for changes in MADRS score) or with non-parametric analysis of two-way ordinal data with repeated measurements34 (for ordinal data). Cognitive data and biological samples will be analysed with t-tests (paired or unpaired as appropriate) or with analysis of variance ANOVA.

Study sample size was calculated based on actual or assumed remission rates, the primary outcome parameter of the study. A remission rate of 60% was set for the reference treatment (ECT). A non-inferiority limit of 40% was set for the experimental intervention (ketamine). This is an arbitrary level, based on an assumption of fewer and milder side effects, faster antidepressant effect and the fact that the patients do not need to be anaesthetized and given muscle relaxants. With the above limits, a power of 80% and a significance level of 5%, 97 patients are required in each arm, according to: n = (2 * 8,4 * p(1-p) / difference2), where "2" and "8,4" are derived from significance and power levels, p are the (actual and assumed) levels for the proportion of patients reaching remission for ECT and ketamine (60% and 40% respectively). The size of the cohort is calculated to be sufficiently large to detect ECT-associated cognitive side effects.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-85
* Diagnosed with major depressive disorder (MDD, according to DSM-IV)
* Inpatients who have been offered and have accepted ECT
* Are eligible to participate
* Score ≥ 20 Points on Montgomery Åsberg Depression Rating Scale (MADRS)
* Must be proficient in spoken and written Swedish
* American Society of Anaesthesiologists physical status classification (ASA) 1-3

Exclusion Criteria:

* Co-morbid conditions that could interfere with the treatment (e.g. primary psychosis)
* Habitual difficulties to speak, hear, remember or reason
* Treatment according to LPT (Lagen om psykiatrisk tvångsvård; Compulsory Psychiatric Care Act)
* On-going or recent (6 months) drug abuse
* Known allergy to the active substance
* Pregnant or breastfeeding women
* Known cardiovascular disease, including angina, acute/chronic congestive heart failure, moderly hypertension or tachyarrhythmia (because exacerbation by sympathomimetic properties of ketamine)
* Pathological conditions in central nervous system with risk of increased intracranial pressure (increased ICP with ketamine)
* Glaucoma (increased IOP with ketamine)
* Porphyria or thyroid disorder (enhanced sympathomimetic properties by ketamine)
* Ongoing severe infection

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2015-02 (Actual); Primary Completion 2019-08 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Proportion of patients in remission in each treatment arm assessed by Montgomery-Asberg Depression Rating Scale (MADRS) | Follow up of one year after treatment cessation
  Primary outcome is the proportion of patients in remission in each treatment arm. Remission is defined as a MADRS ≤ 10.

SECONDARY OUTCOMES:
Time to remission compared between the two treatments. | The MADRS score is measured for a maximum of 4 weeks.
  Time (days) to reach remission (defined as MADRS≤ 10) is compared between the groups.
Time to response compared between the two treatments. | The MADRS score is measured for a maximum of 4 weeks.
  Time (days) to response (defined as a drop of 50% from the pre-treatment MADRS value)) is compared between the groups.
Ketamine treatment is associated with a smaller decrease in the performance in a CANTAB cognitive test battery compared to ECT. | Assessed prior to the first treatment, after two weeks, within one week after remission and at three additional time points (3, 6 and 12 months) after conclusion of the treatment.
  Cognitive function are assessed with Cambridge Automated Neuropsychological Test Automated Battery (CANTAB).
Remission from severe depression is associated with improved performance in the performance in a CANTAB cognitive test battery. | Assessed prior to the first treatment, after two weeks, within one week after remission and at three additional time points (3, 6 and 12 months) after conclusion of the treatment.
  Cognitive function are assessed with Cambridge Automated Neuropsychological Test Automated Battery (CANTAB).
The antidepressant effect of ketamine is longer lasting than that of ECT, assessed by the proportion of patients in remission (defined by a maximum score of 9 in the Montgomery-Asberg Depression Rating Scale (MADRS)). | Within one week after remission and at three additional time points (3, 6 and 12 months) after remission
  The antidepressant effect will be assessed with MADRS baseline score and measured within one week after remission and at three additional time points (3, 6 and 12 months) after conclusion of the treatment.
Ketamine treatment is associated with a smaller decrease in the performance in Rey Auditory Verbal Learning Test (RAVLT) compared to ECT. | Assessed prior to the first treatment, after two weeks, within one week after remission and at three additional time points (3, 6 and 12 months) after conclusion of the treatment.
  Reys Auditory Verbal Learning Test (RAVLT)
Remission from severe depression is associated with improved performance in the performance in Rey Auditory Verbal Learning Test (RAVLT). | Assessed prior to the first treatment, after two weeks, within one week after remission and at three additional time points (3, 6 and 12 months) after conclusion of the treatment.
  Reys Auditory Verbal Learning Test (RAVLT)

CONTACTS AND LOCATIONS:
Overall Officials: Pouya Movahed Rad, MD, PhD, Principal Investigator — Dept of Clinical Sciences Lund, Faculty of Medicine Lund University, Sweden
Locations (1):
- Department of Psychiatry, Lund, Sweden

IPD SHARING:
Plan to Share IPD: Undecided